CLINICAL TRIAL: NCT06211517
Title: Subjective Experience of Psychotropic Drugs Among Adolescents (Their Parents and Professionals) With Anorexia Nervosa
Brief Title: Drugs Experience for Adolescents With Anorexia
Acronym: E3P
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230062; 2022-A02141-42 (Other: France : Ministry of Health)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Anorexia Nervosa; Psychotropic Drugs; Adolescent
Keywords: Adolescents; Anorexia nervosa; Psychotropic drugs; Qualitative research; Thematic analysis
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Adolescents: Adolescents suffering from anorexia nervosa 12 to 25 years
  Interventions: Other: Semi-structured interviews with visual mediations
- Parents: Parents whose adolescents suffer from anorexia nervosa
  Interventions: Other: Semi-structured interviews with visual mediations
- Healthcare professionals: Healthcare professionals in charge of adolescents suffering from anorexia nervosa
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews with visual mediations — Semi-structured interviews with visual mediations / An hour-long interview
  Other Names: Qualitative interviews
  Groups: Adolescents; Parents
Other: Semi-structured interviews — Semi-structured interviews
  Other Names: Qualitative interviews
  Groups: Healthcare professionals

SUMMARY:
The purpose of this study is to access to the experiences of adolescents, their parents and healthcare professionals regarding psychotropic drugs in anorexia nervosa.

No preconceived ideas (according to qualitative methods) but a question: what are the participants' perceptions and experiences of psychotropic drugs in anorexia nervosa? In an adolescent medicine department.

DETAILED DESCRIPTION:
Psychotropic prescription is common to adolescents suffering from anorexia nervosa. A first qualitative study (E3A Protocol "Experience of adolescents with anorexia nervosa toward antidepressants") looked at the experience of antidepressants among 15 adolescents suffering from anorexia nervosa. Analysis of the interviews identified two meta-themes:

1. Reactions to the proposal of antidepressant with an opposition phase (about the existence of depressive symptoms and about negative preconceptions) and need to share with family and other teenagers.
2. Reactions to antidepressant use with ambivalence and an initial perception of coercion, and effects of antidepressants (psychological effects, effects on the body and on anorexia nervosa and effects perceived through the eyes of others).

Nine adolescents (out of 15) were also taking an atypical antipsychotic (APA) often prescribed in case of anorexia nervosa resistance.

The need to share with family about the proposal of antidepressant and the effects perceived through the eyes of others (including parent's eyes) lead us to take an interest in parents perceptions.

Two decisive periods were identified: What do healthcare professionals think about psychotropic treatments for anorexia nervosa in adolescence? How do they propose treatment?

Interviewing teenagers, their parents as well as healthcare professionals, will enable to access to the complexity of representations and experiences of these psychotropic drugs in anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

Adolescents :

* Aged 12 to 25 years
* Suffering from anorexia nervosa (restrictive or mixed) according to DSM-5 (Diagnostic and Statistical Manual) criteria
* Received psychotropic drugs (antidepressant treatment and/or APA) during their care, either ongoing or discontinued before this study started

Parents of adolescents suffering from anorexia nervosa for whom a psychotropic drug has been prescribed and whose adolescents meet inclusion criteria

Healthcare Professionals working with adolescents suffering from eating disorders

Exclusion Criteria:

Adolescents :

* Atypical eating disorder that does not meet the DSM-5 criteria for restrictive or mixed anorexia nervosa
* BMI<15
* Prescription of an antidepressant other than an SSRI (Selective Serotonin Reuptake Inhibitor)
* Prescription of an APA for the indication of psychotic symptoms

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent medicine department in Cochin hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Semi-structured interview | Day of inclusion
  Themes describing adolescent experiences regarding psychotropic drugs in anorexia nervosa - Emergence of themes describing participants' experience from analysis of qualitative interviews (with Interpretative Phenomenology Analysis methodology)

SECONDARY OUTCOMES:
Semi-structured interview | Day of inclusion
  Themes describing parents experiences regarding psychotropic drugs for their children suffering from anorexia nervosa - Emergence of themes describing participants' experience from analysis of qualitative interviews (with Interpretative Phenomenology Analysis methodology)
Semi-structured interview | Day of inclusion
  Themes describing healthcare professionals experiences regarding psychotropic drugs for adolescents suffering from anorexia nervosa - Emergence of themes describing participants' experience from analysis of qualitative interviews (with Interpretative Phenomenology Analysis methodology)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Blanchet, MD, Study Director — Cochin Hospital (maison de Solenn); Marie Rose Moro, MD, PhD, Study Director — Cochin Hospital (maison de Solenn); Maude Ludot-Gregoire, MD, Principal Investigator — Cochin Hospital (maison de Solenn)
Locations (1):
- Maison de Solenn Maison des Adolescents, Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ludot-Gregoire M, David V, Carretier E, Lachal J, Moro MR, Blanchet C. Subjective Experience of Antidepressant Prescription Among Adolescents With Anorexia Nervosa. Front Psychiatry. 2022 Apr 4;13:770903. doi: 10.3389/fpsyt.2022.770903. eCollection 2022. PMID 35444576
- See also: First qualitative study (E3A Protocol) — https://doi.org/10.3389/fpsyt.2022.770903